CLINICAL TRIAL: NCT00695266
Title: Profile of Hypertensive Patients Seen in Hospital Outpatient's Department
Brief Title: National Survey on Hypertension at Hospital
Acronym: PROPHYL HO
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Alain Castaigne, Medical Director, AstraZeneca Pharmaceuticals
Other Study IDs: NIS-CFR-DUM-2007/5
Record Dates: First submitted 2008-06-09; First posted 2008-06-11 (Estimated); Last update posted 2009-08-06 (Estimated); Status verified 2009-08

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1

SUMMARY:
To evaluate (with sufficient accuracy) the profile(demographic and clinical characteristics, health care management) of hypertensive patients seen in hospital out patient's department by a cardiologist or a nephrologists.

ELIGIBILITY:
Inclusion Criteria:

* Known hypertension
* agree to take part in this study

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: First five consecutive patients with hypertension seen by Cardiologists
Sampling Method: Probability Sample
Enrollment: 655 (Actual)
Dates: Start 2007-12; Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Demographic, clinical and health care characteristics | Once

CONTACTS AND LOCATIONS:
Locations (113):
- France (113):
  - Research Site, Abreschviller
  - Research Site, Aix-en-Provence
  - Research Site, Ajaccio
  - Research Site, Ambilly
  - Research Site, Annecy
  - Research Site, Auch
  - Research Site, Auxerre
  - Research Site, Bar-le-Duc
  - Research Site, Bastia
  - Research Site, Bobigny
  - Research Site, Bourges
  - Research Site, Bron
  - Research Site, Bry-sur-Marne
  - Research Site, Cahors
  - Research Site, Caluire-et-Cuire
  - Research Site, Cambo-les-Bains
  - Research Site, Cambrai
  - Research Site, Chalon-sur-Saône
  - Research Site, Chambéry
  - Research Site, Chambray-lès-Tours
  - Research Site, Champigny-sur-Marne
  - Research Site, Charleville-Mézières
  - Research Site, Chaumont
  - Research Site, Chauny
  - Research Site, Châteauroux
  - Research Site, Cholet
  - Research Site, Colmar
  - Research Site, Corbeil-Essonnes
  - Research Site, Creil
  - Research Site, Créteil
  - Research Site, Dax
  - Research Site, Dechy
  - Research Site, Décines-Charpieu
  - Research Site, Dieppe
  - Research Site, Dijon
  - Research Site, Dunkirk
  - Research Site, Eaubonne
  - Research Site, Évecquemont
  - Research Site, Évian-les-Bains
  - Research Site, Firminy
  - Research Site, Forbach
  - Research Site, Freyming-Merlebach
  - Research Site, Gap
  - Research Site, Givors
  - Research Site, Gleizé
  - Research Site, Gonesse
  - Research Site, Grenoble
  - Research Site, Haguenau
  - Research Site, Hyères
  - Research Site, La Rochelle
  - Research Site, La Source
  - Research Site, Lagny-sur-Marne
  - Research Site, Langres
  - Research Site, Lannion
  - Research Site, Laon
  - Research Site, Laval
  - Research Site, Le Chesnay
  - Research Site, Le Puy-en-Velay
  - Research Site, Libourne
  - Research Site, Limoges
  - Research Site, Lunéville
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Martigues
  - Research Site, Melun
  - Research Site, Metz
  - Research Site, Mont-de-Marsan
  - Research Site, Montfermeil
  - Research Site, Montivilliers
  - Research Site, Montpellier
  - Research Site, Montreuil
  - Research Site, Nice
  - Research Site, Niort
  - Research Site, Nîmes
  - Research Site, Orange
  - Research Site, Oyonnax
  - Research Site, Paray-le-Monial
  - Research Site, Paris
  - Research Site, Pau
  - Research Site, Pessac
  - Research Site, Périgueux
  - Research Site, Pierre-Bénite
  - Research Site, Poissy
  - Research Site, Pontault-Combault
  - Research Site, Provins
  - Research Site, Roanne
  - Research Site, Saint-Amand-Montrond
  - Research Site, Saint-Avold
  - Research Site, Saint-Herblain
  - Research Site, Saint-Martin-d'Aubigny
  - Research Site, Saint-Priest-en-Jarez
  - Research Site, Saint-Quentin
  - Research Site, Sallanches
  - Research Site, Salouël
  - Research Site, Sarreguemines
  - Research Site, Schiltigheim
  - Research Site, Semur-en-Auxois
  - Research Site, Senlis
  - Research Site, Sisteron
  - Research Site, Strasbourg
  - Research Site, Suresnes
  - Research Site, Tarbes
  - Research Site, Thiais
  - Research Site, Toulon Armees
  - Research Site, Toulouse
  - Research Site, Tours
  - Research Site, Tracy-le-Mont
  - Research Site, Trappes
  - Research Site, Tulle
  - Research Site, Vandœuvre-lès-Nancy
  - Research Site, Vénissieux
  - Research Site, Villenave-d'Ornon
  - Research Site, Villeneuve-Saint-Georges